CLINICAL TRIAL: NCT01379469
Title: A Preliminary Study of the Efficacy and Safety of Carbamazepine in Severe Liver Disease Due to Alpha-1 Antitrypsin Deficiency
Brief Title: Carbamazepine in Severe Liver Disease Due to Alpha-1 Antitrypsin Deficiency
Acronym: CBZ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis (Industry); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201510060-PRO09070279; 1R21DK092567-01 (NIH)
Record Dates: First submitted 2011-06-15; First posted 2011-06-23 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Alpha-1-antitrypsin Deficiency; Liver Cirrhosis
Keywords: Carbamazepine (Tegretol) use; severe liver disease; alpha-1-antitrypsin deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Liver Cirrhosis; Liver Diseases | interventions — Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug-Carbamazepine (Tegretol XR) (Active Comparator): One arm receives Drug-Carbamazepine (Tegretol XR).All subjects have severe liver disease due to alpha-1-antitrypsin deficiency.
  Interventions: Drug: Drug-Carbamazepine (Tegretol XR)
- Drug-Carbamazepine (Tegretol XR) Placebo (Placebo Comparator): One arm receives Carbamazepine (Tegretol-XR) placebo.All subjects have severe liver disease due to alpha-1-antitrypsin deficiency.
  Interventions: Drug: Carbamazepine (Tegretol XR) Placebo

INTERVENTIONS:
Drug: Drug-Carbamazepine (Tegretol XR) — To reduce the likelihood of hypersensitivity reactions the subjects will be started on 400 mg/day in 2 doses and the dose will be increased weekly by 200mg/day until reaching a stable therapeutic concentration with a dose not exceeding 1200mg/day(or 1000mg/day in subjects less than 15 years of age). The CBZ tablets will be encapsulated..
  Other Names: Tegretol-XR Carbamazepine extended release tablets.; NDC 0078-0510-05.
  Arms: Drug-Carbamazepine (Tegretol XR)
Drug: Carbamazepine (Tegretol XR) Placebo — Carbamazepine (Tegretol XR)Placebo-the subjects will be started on 400mg/day in 2 doses and the dose will be increased weekly by 200 mg/day until reaching a dose not exceeding 1200 mg/day (or 1000 mg/day in subjects less than 15 years of age). The placebo group will receive encapsulated tables without Carbamazepine.
  Other Names: Carbamazepine (Tegretol-XR) placebo.
  Arms: Drug-Carbamazepine (Tegretol XR) Placebo

SUMMARY:
The primary objective is to determine if the medication Carbamazepine, can be used as a therapy for patients with severe liver disease due to Alpha-1-Antitrypsin Deficiency .

DETAILED DESCRIPTION:
The primary objective is to determine if Carbamazepine therapy in patients with severe liver disease due to Alpha-1-Antitrypsin Deficiency leads to a significant reduction in the hepatic accumulation of ATZ.

The other objectives are:

To determine whether Carbamazepine treatment reduces hepatic fibrosis in alpha-1-antitrypsin deficient patients with severe liver disease. To determine whether Carbamazepine treatment reduces portal pressure in alpha-1-antitrypsin deficient patients with severe liver disease. To determine whether Carbamazepine treatment is safe and tolerated by patients with severe liver disease caused by alpha-1-deficiency. To determine whether Carbamazepine treatment leads to stabilization in disease severity as measured by the MELD scores.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 14 years to less than or equal to 80 years of age.
* Alpha-1-Antitrypsin deficiency confirmed by ZZ or SZ phenotype & serum level
* < 83mg/dl.
* HVPG greater than or equal to 10 mmHg unless collateral vessels are visualized via transvenous biopsy.

Exclusion Criteria:

* Child Pugh Score greater than or equal to 12. Serum total bilirubin > 5 mg/dl. INR > 2.2.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Perlmutter, M.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Children's Hospital of Pittsburgh, UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Presbyterian Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We will share data and liver tissue with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. We may also share research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at the information.

REFERENCES:
- [Background] Perlmutter D.H., Alpha-1-Antitrypsin Deficiency, in Schiff's Disease of Liver, Schiff E.R., Maddrey W.C., Editor. 2007; Lippincott-Raven: Philadelphia. 1063-1084.
- [Background] Perlmutter DH. Pathogenesis of chronic liver injury and hepatocellular carcinoma in alpha-1-antitrypsin deficiency. Pediatr Res. 2006 Aug;60(2):233-8. doi: 10.1203/01.pdr.0000228350.61496.90. PMID 16864711
- [Background] Perlmutter DH. Autophagic disposal of the aggregation-prone protein that causes liver inflammation and carcinogenesis in alpha-1-antitrypsin deficiency. Cell Death Differ. 2009 Jan;16(1):39-45. doi: 10.1038/cdd.2008.103. Epub 2008 Jul 11. PMID 18617899
- [Background] Rudnick DA, Perlmutter DH. Alpha-1-antitrypsin deficiency: a new paradigm for hepatocellular carcinoma in genetic liver disease. Hepatology. 2005 Sep;42(3):514-21. doi: 10.1002/hep.20815. PMID 16044402
- [Background] Piitulainen E, Carlson J, Ohlsson K, Sveger T. Alpha1-antitrypsin deficiency in 26-year-old subjects: lung, liver, and protease/protease inhibitor studies. Chest. 2005 Oct;128(4):2076-81. doi: 10.1378/chest.128.4.2076. PMID 16236857
- [Background] Sveger T. Liver disease in alpha1-antitrypsin deficiency detected by screening of 200,000 infants. N Engl J Med. 1976 Jun 10;294(24):1316-21. doi: 10.1056/NEJM197606102942404. PMID 1083485
- [Background] Eriksson S, Carlson J, Velez R. Risk of cirrhosis and primary liver cancer in alpha 1-antitrypsin deficiency. N Engl J Med. 1986 Mar 20;314(12):736-9. doi: 10.1056/NEJM198603203141202. PMID 3485248
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913
- [Background] Malinchoc M, Kamath PS, Gordon FD, Peine CJ, Rank J, ter Borg PC. A model to predict poor survival in patients undergoing transjugular intrahepatic portosystemic shunts. Hepatology. 2000 Apr;31(4):864-71. doi: 10.1053/he.2000.5852. PMID 10733541
- [Background] Burroughs AK, Thalheimer U. Hepatic venous pressure gradient in 2010: optimal measurement is key. Hepatology. 2010 Jun;51(6):1894-6. doi: 10.1002/hep.23710. No abstract available. PMID 20512984
- [Background] Zoli M, Iervese T, Merkel C, Bianchi G, Magalotti D, Marchesini G, Gatta A, Pisi E. Prognostic significance of portal hemodynamics in patients with compensated cirrhosis. J Hepatol. 1993 Jan;17(1):56-61. doi: 10.1016/s0168-8278(05)80521-5. PMID 8445220
- [Background] Manolakopoulos S, Triantos C, Theodoropoulos J, Vlachogiannakos J, Kougioumtzan A, Papatheodoridis G, Tzourmakliotis D, Karamanolis D, Burroughs AK, Archimandritis A, Raptis S, Avgerinos A. Antiviral therapy reduces portal pressure in patients with cirrhosis due to HBeAg-negative chronic hepatitis B and significant portal hypertension. J Hepatol. 2009 Sep;51(3):468-74. doi: 10.1016/j.jhep.2009.05.031. Epub 2009 Jul 3. PMID 19616339
- [Background] Roberts S, Gordon A, McLean C, Pedersen J, Bowden S, Thomson K, Angus P. Effect of sustained viral response on hepatic venous pressure gradient in hepatitis C-related cirrhosis. Clin Gastroenterol Hepatol. 2007 Aug;5(8):932-7. doi: 10.1016/j.cgh.2007.02.022. Epub 2007 Jun 4. PMID 17544878
- [Background] Hidvegi T., Perlmutter D.H., Watkins S., and Michalopoulos G., Carbamazepine ameliorates liver disease in mouse models of alpha-1-antitrypsin deficiency by enhancing intracellular disposal of the pathogenic aggregation-prone protein. Science; 2010; 329: 229-232.
- [Background] Dodson W., Carbamazepine and oxycarbazepine, Pediatric Epilepsy: Diagnosis and Therapy, P.J. Dodson W.E., Editor. 1993; Demos Publications: New York. 303-314.
- [Background] Williams RS, Cheng L, Mudge AW, Harwood AJ. A common mechanism of action for three mood-stabilizing drugs. Nature. 2002 May 16;417(6886):292-5. doi: 10.1038/417292a. PMID 12015604
- [Background] Sarkar S, Floto RA, Berger Z, Imarisio S, Cordenier A, Pasco M, Cook LJ, Rubinsztein DC. Lithium induces autophagy by inhibiting inositol monophosphatase. J Cell Biol. 2005 Sep 26;170(7):1101-11. doi: 10.1083/jcb.200504035. PMID 16186256
- [Background] McNamara J., Drugs effective in the therapy of epilepsies, Goodman and Gillman's: The Pharmacological Basis of Therapeutics, J. Hardman, L. Limbird, and A. Cillman, Editors. 2001; McGraw-Hill: New York. 533-535.
- [Background] Wada JA, Troupin AS, Friel P, Remick R, Leal K, Pearmain J. Pharmacokinetic comparison of tablet and suspension dosage forms of carbamazepine. Epilepsia. 1978 Jun;19(3):251-5. doi: 10.1111/j.1528-1157.1978.tb04487.x. PMID 679894
- [Background] Chung WH, Hung SI, Hong HS, Hsih MS, Yang LC, Ho HC, Wu JY, Chen YT. Medical genetics: a marker for Stevens-Johnson syndrome. Nature. 2004 Apr 1;428(6982):486. doi: 10.1038/428486a. PMID 15057820
- [Background] Man CB, Kwan P, Baum L, Yu E, Lau KM, Cheng AS, Ng MH. Association between HLA-B*1502 allele and antiepileptic drug-induced cutaneous reactions in Han Chinese. Epilepsia. 2007 May;48(5):1015-8. doi: 10.1111/j.1528-1167.2007.01022.x. Erratum In: Epilepsia. 2008 May;49(5):941. PMID 17509004
- [Background] McCormack M, Alfirevic A, Bourgeois S, Farrell JJ, Kasperaviciute D, Carrington M, Sills GJ, Marson T, Jia X, de Bakker PI, Chinthapalli K, Molokhia M, Johnson MR, O'Connor GD, Chaila E, Alhusaini S, Shianna KV, Radtke RA, Heinzen EL, Walley N, Pandolfo M, Pichler W, Park BK, Depondt C, Sisodiya SM, Goldstein DB, Deloukas P, Delanty N, Cavalleri GL, Pirmohamed M. HLA-A*3101 and carbamazepine-induced hypersensitivity reactions in Europeans. N Engl J Med. 2011 Mar 24;364(12):1134-43. doi: 10.1056/NEJMoa1013297. PMID 21428769
- [Background] Chen P, Lin JJ, Lu CS, Ong CT, Hsieh PF, Yang CC, Tai CT, Wu SL, Lu CH, Hsu YC, Yu HY, Ro LS, Lu CT, Chu CC, Tsai JJ, Su YH, Lan SH, Sung SF, Lin SY, Chuang HP, Huang LC, Chen YJ, Tsai PJ, Liao HT, Lin YH, Chen CH, Chung WH, Hung SI, Wu JY, Chang CF, Chen L, Chen YT, Shen CY; Taiwan SJS Consortium. Carbamazepine-induced toxic effects and HLA-B*1502 screening in Taiwan. N Engl J Med. 2011 Mar 24;364(12):1126-33. doi: 10.1056/NEJMoa1009717. PMID 21428768
- [Background] Vigo DV, Baldessarini RJ. Anticonvulsants in the treatment of major depressive disorder: an overview. Harv Rev Psychiatry. 2009;17(4):231-41. doi: 10.1080/10673220903129814. PMID 19637072
- [Background] Huband N, Ferriter M, Nathan R, Jones H. Antiepileptics for aggression and associated impulsivity. Cochrane Database Syst Rev. 2010 Feb 17;2010(2):CD003499. doi: 10.1002/14651858.CD003499.pub3. PMID 20166067
- [Background] Minozzi S, Amato L, Vecchi S, Davoli M. Anticonvulsants for alcohol withdrawal. Cochrane Database Syst Rev. 2010 Mar 17;2010(3):CD005064. doi: 10.1002/14651858.CD005064.pub3. PMID 20238337
- [Background] Zakrzewska JM. Medical management of trigeminal neuropathic pains. Expert Opin Pharmacother. 2010 Jun;11(8):1239-54. doi: 10.1517/14656561003767449. PMID 20426709
- [Background] Wilkinson GR, Schenker S. Drug disposition and liver disease. Drug Metab Rev. 1975;4(2):139-75. doi: 10.3109/03602537508993754. No abstract available. PMID 770104
- [Background] Mueller TI, Stout RL, Rudden S, Brown RA, Gordon A, Solomon DA, Recupero PR. A double-blind, placebo-controlled pilot study of carbamazepine for the treatment of alcohol dependence. Alcohol Clin Exp Res. 1997 Feb;21(1):86-92. PMID 9046378
- [Background] Clark JM, Brancati FL, Diehl AM. The prevalence and etiology of elevated aminotransferase levels in the United States. Am J Gastroenterol. 2003 May;98(5):960-7. doi: 10.1111/j.1572-0241.2003.07486.x. PMID 12809815
- [Background] Tandra S, Vuppalanchi R. Use of statins in patients with liver disease. Curr Treat Options Cardiovasc Med. 2009 Aug;11(4):272-8. doi: 10.1007/s11936-009-0028-2. PMID 19627660
- [Background] Ishizu H, Shiomi S, Kawamura E, Iwata Y, Nishiguchi S, Kawabe J, Ochi H. Gastric emptying in patients with chronic liver diseases. Ann Nucl Med. 2002 May;16(3):177-82. doi: 10.1007/BF02996298. PMID 12126042
- [Background] Parlesak A, Schafer C, Schutz T, Bode JC, Bode C. Increased intestinal permeability to macromolecules and endotoxemia in patients with chronic alcohol abuse in different stages of alcohol-induced liver disease. J Hepatol. 2000 May;32(5):742-7. doi: 10.1016/s0168-8278(00)80242-1. PMID 10845660
- [Background] Morgan DJ, McLean AJ. Clinical pharmacokinetic and pharmacodynamic considerations in patients with liver disease. An update. Clin Pharmacokinet. 1995 Nov;29(5):370-91. doi: 10.2165/00003088-199529050-00005. PMID 8582120
- [Background] Verbeeck RK, Horsmans Y. Effect of hepatic insufficiency on pharmacokinetics and drug dosing. Pharm World Sci. 1998 Oct;20(5):183-92. doi: 10.1023/a:1008656930082. PMID 9820880
- [Background] Rodriquez A, Martin A, Oterino JA, Blanco I, Jimenez M, Perez A, Novoa JM. Renal function in compensated hepatic cirrhosis: effects of an amino acid infusion and relationship with nitric acid. Dig Dis. 1999;17(4):235-40. doi: 10.1159/000016942. PMID 10754364
- [Background] Delco F, Tchambaz L, Schlienger R, Drewe J, Krahenbuhl S. Dose adjustment in patients with liver disease. Drug Saf. 2005;28(6):529-45. doi: 10.2165/00002018-200528060-00005. PMID 15924505
- [Background] George J, Liddle C, Murray M, Byth K, Farrell GC. Pre-translational regulation of cytochrome P450 genes is responsible for disease-specific changes of individual P450 enzymes among patients with cirrhosis. Biochem Pharmacol. 1995 Mar 30;49(7):873-81. doi: 10.1016/0006-2952(94)00515-n. PMID 7741759
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Cholongitas E, Senzolo M, Standish R, Marelli L, Quaglia A, Patch D, Dhillon AP, Burroughs AK. A systematic review of the quality of liver biopsy specimens. Am J Clin Pathol. 2006 May;125(5):710-21. doi: 10.1309/W3XC-NT4H-KFBN-2G0B. PMID 16707372
- [Background] Kalambokis G, Manousou P, Vibhakorn S, Marelli L, Cholongitas E, Senzolo M, Patch D, Burroughs AK. Transjugular liver biopsy--indications, adequacy, quality of specimens, and complications--a systematic review. J Hepatol. 2007 Aug;47(2):284-94. doi: 10.1016/j.jhep.2007.05.001. Epub 2007 May 24. PMID 17561303
- [Background] Vibhakorn S, Cholongitas E, Kalambokis G, Manousou P, Quaglia A, Marelli L, Senzolo M, Patch D, Dhillon A, Burroughs AK. A comparison of four- versus three-pass transjugular biopsy using a 19-G Tru-Cut needle and a randomized study using a cassette to prevent biopsy fragmentation. Cardiovasc Intervent Radiol. 2009 May;32(3):508-13. doi: 10.1007/s00270-008-9412-7. Epub 2008 Aug 13. PMID 18704569
- [Background] Miller AD, Krauss GL, Hamzeh FM. Improved CNS tolerability following conversion from immediate- to extended-release carbamazepine. Acta Neurol Scand. 2004 Jun;109(6):374-7. doi: 10.1111/j.1600-0404.2004.00291.x. PMID 15147458
- [Background] Brent DA, Emslie GJ, Clarke GN, Asarnow J, Spirito A, Ritz L, Vitiello B, Iyengar S, Birmaher B, Ryan ND, Zelazny J, Onorato M, Kennard B, Mayes TL, Debar LL, McCracken JT, Strober M, Suddath R, Leonard H, Porta G, Keller MB. Predictors of spontaneous and systematically assessed suicidal adverse events in the treatment of SSRI-resistant depression in adolescents (TORDIA) study. Am J Psychiatry. 2009 Apr;166(4):418-26. doi: 10.1176/appi.ajp.2008.08070976. Epub 2009 Feb 17. PMID 19223438
- [Background] Emslie GJ, Mayes T, Porta G, Vitiello B, Clarke G, Wagner KD, Asarnow JR, Spirito A, Birmaher B, Ryan N, Kennard B, DeBar L, McCracken J, Strober M, Onorato M, Zelazny J, Keller M, Iyengar S, Brent D. Treatment of Resistant Depression in Adolescents (TORDIA): week 24 outcomes. Am J Psychiatry. 2010 Jul;167(7):782-91. doi: 10.1176/appi.ajp.2010.09040552. Epub 2010 May 17. PMID 20478877
- [Background] Shemesh E, Shneider BL, Savitzky JK, Arnott L, Gondolesi GE, Krieger NR, Kerkar N, Magid MS, Stuber ML, Schmeidler J, Yehuda R, Emre S. Medication adherence in pediatric and adolescent liver transplant recipients. Pediatrics. 2004 Apr;113(4):825-32. doi: 10.1542/peds.113.4.825. PMID 15060234
- [Background] Frey B, Schubiger G, Musy JP. Transient cholestatic hepatitis in a neonate associated with carbamazepine exposure during pregnancy and breast-feeding. Eur J Pediatr. 1990 Dec;150(2):136-8. doi: 10.1007/BF02072057. PMID 2279511
- [Derived] Silverman GA, Pak SC, Perlmutter DH. Disorders of protein misfolding: alpha-1-antitrypsin deficiency as prototype. J Pediatr. 2013 Aug;163(2):320-6. doi: 10.1016/j.jpeds.2013.03.077. Epub 2013 May 8. No abstract available. PMID 23664631

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug-Carbamazepine (Tegretol XR) | Drug-Carbamazepine (Tegretol XR) Placebo
Started | 13 | 7
Completed | 1 | 3
Not Completed | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Drug-Carbamazepine (Tegretol XR): One arm receives Drug-Carbamazepine (Tegretol XR).All subjects have severe liver disease due to alpha-1-antitrypsin deficiency.
  Drug-Carbamazepine (Tegretol XR): To reduce the likelihood of hypersensitivity reactions the subjects will be started on 400 mg/day in 2 doses and the dose will be increased weekly by 200mg/day until reaching a stable therapeutic concentration with a dose not exceeding 1200mg/day(or 1000mg/day in subjects less than 15 years of age). The CBZ tablets will be encapsulated, and the placebo group will receive encapsulated tablets without CBZ.
- Total: Total of all reporting groups
Arm/Group | Drug-Carbamazepine (Tegretol XR) | Drug-Carbamazepine (Tegretol XR) Placebo | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 13 | 3 | 16
  >=65 years | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (9.4) | 53.7 (19.6) | 51.75 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 8 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 7 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be to Determine the Effect of Carbamazepine on Hepatic ATZ Load.
Description: The effect of Carbamazepine on hepatic ATZ load will be measured by the number of hepatocytes with PAS+/diastase-resistant globules and/or steady state levels of ATZ by immunoblot analysis.
Time Frame: 52 weeks
Population: The primary outcome was not assessable because the number of subjects with available pre & post PAS+/diastase stained liver biopsies & tissue for immunoblot was insufficient in subject number and sample quality. To elaborate only 3 subjects had both pre & post biopsies stained for PAS, 2 from the placebo & 1 from the Carbamazepine arms & the available histology quality was insufficient for histomorphormetry. Frozen liver samples were also of insufficient number & mass for immunoblot.
Arm/Group | Drug-Carbamazepine (Tegretol XR) | Drug-Carbamazepine (Tegretol XR) Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: For the Secondary Outcomes we Will Determine the Effect of Carbamazepine Treatment on Hepatic Fibrosis.
Description: For the secondary outcomes we will determine the effect of Carbamazepine treatment on hepatic fibrosis on the basis of sirius red staining and hydroxyproline concentration and whether Carbamazepine treatment changes portal pressure as determined by Hepatic Venous Pressure Gradient.
Time Frame: 52 weeks
Population: The secondary outcome was also not assessable because the number of subjects with available pre & post trichrome stained liver biopsies & tissue for hydroxyproline was also insufficient in subject number and sample quality. Again only 3 subjects had both pre & post biopsies stained for trichrome, 2 placebo- & 1 Carbamazepine treated. Available histology quality was also insufficient here for histomorphormetry &.frozen liver samples insufficient for hydroxyproline determination.
Arm/Group | Drug-Carbamazepine (Tegretol XR) | Drug-Carbamazepine (Tegretol XR) Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Adverse Events were collected for 52 weeks.
Arm/Group | Drug-Carbamazepine (Tegretol XR) | Drug-Carbamazepine (Tegretol XR) Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 2/7
Serious Adverse Events (participants affected / at risk) | 6/13 | 4/7
Other Adverse Events (participants affected / at risk) | 13/13 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-Carbamazepine (Tegretol XR) (N=13) | Drug-Carbamazepine (Tegretol XR) Placebo (N=7)
Gastrointestinal (Gastrointestinal disorders) | 2 (3) | 2 (2)
Pain (General disorders) | 2 (3) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Cardiac (Cardiac disorders) | 1 (1) | 1 (2)
Infection (Infections and infestations) | 2 (4) | 2 (2)
Vascular (Vascular disorders) | 2 (2) | 0 (0)
Constitutional (General disorders) | 4 (6) | 0 (0)
Hematologic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-Carbamazepine (Tegretol XR) (N=13) | Drug-Carbamazepine (Tegretol XR) Placebo (N=7)
Cardiac (Cardiac disorders) | 1 (2) | 3 (4)
Child-Pugh Score Increase (Hepatobiliary disorders) | 1 (1) | 1 (2)
Constitutional (General disorders) | 12 (63) | 7 (17)
Dermatologic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4)
Endocrine (Endocrine disorders) | 3 (3) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 9 (35) | 5 (13)
Genitourological (Renal and urinary disorders) | 3 (3) | 2 (2)
Gynecological (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Hematologic (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Infection (Infections and infestations) | 7 (16) | 3 (5)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 (12) | 3 (5)
Neurologic (Nervous system disorders) | 10 (31) | 3 (5)
Pain (General disorders) | 8 (15) | 5 (8)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 4 (5)
Vascular (Vascular disorders) | 5 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary & secondary outcomes could not be assessed because the number of subjects with available pre & post biopsies was insufficient in subject number and sample quality to conduct the analyses. As described in more detail in Outcome Measures.

.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT01379469/Prot_SAP_000.pdf